CLINICAL TRIAL: NCT01137435
Title: Regulatory Post-Marketing Surveillance (PMS) Study for ADACEL™ (Adsorbed Diphtheria, Tetanus Toxoids and Component Pertussis Combined Vaccine for Adult)
Brief Title: Post Marketing Surveillance for ADACEL™ in South Korea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Td533; UTN: U1111-1112-8558 (Other: WHO)
Record Dates: First submitted 2010-06-03; First posted 2010-06-04 (Estimated); Results first posted 2017-01-04 (Estimated); Last update posted 2022-04-28 (Actual); Status verified 2022-03

CONDITIONS: Diphtheria; Tetanus; Pertussis
Keywords: Adacel; Diphtheria; Tetanus; Pertussis
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough | interventions — Tetanus Toxoid; adacel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study Group (Experimental)
  Interventions: Biological: ADACEL™:Adsorbed Diphtheria, Tetanus Toxoids and Component Pertussis Combined

INTERVENTIONS:
Biological: ADACEL™:Adsorbed Diphtheria, Tetanus Toxoids and Component Pertussis Combined — 0.5 mL, intramuscular (IM)
  Other Names: Adacel™

SUMMARY:
This safety surveillance study is being conducted in accordance with Korea Food and Drug Administration (KFDA) Notification No. 2009-46 "Basic standard for reexamination of new drug".

The study objective is to assess within 30 days post-administration, the safety of ADACEL™ administered under the real clinical practice.

ELIGIBILITY:
Inclusion Criteria :

* Subjects who are 11 through 64 years of age (as indicated in the currently approved local product labeling) , who are given a single dose of the study vaccine, during a routine health-care visit, as active booster immunization for the prevention of tetanus, diphtheria and pertussis.
* Written informed consent obtained from the subject. For subjects below the legal age of consent, written informed consent must be obtained from the parent or legal guardian (legally acceptable representative -LAR) of the subject.

Exclusion Criteria :

* None

Ages: 11 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 659 (Actual)
Dates: Start 2010-06; Primary Completion 2016-03 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur Inc.
Locations (2):
- South Korea (2):
  - Jung-gu, Incheon
  - Seoul

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Post Marketing Surveillance period was from 23 June 2009 to 22 June 2015 at 7 clinic centers in South Korea.
Pre-assignment Details: Case report forms were retrieved from a total of 687 participants during the 6 years post marketing surveillance study; 659 participants were included in the safety analysis.
Groups:
- Study Subjects: Participants who had returned case report forms and included in the safety analysis.
Period: Overall Study
Arm/Group | Study Subjects
Started | 687
Completed | 659
Not Completed | 28
Not completed — Lost to Follow-up | 24
Not completed — Off label usage | 4

BASELINE CHARACTERISTICS:
Arm/Group | Study Subjects
Number analyzed (Participants) | 659
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 275
  Between 18 and 65 years | 384
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 24.38 (13.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 454
  Male | 205
Region of Enrollment [Number; unit: Participants]
  Korea, Republic of | 659

OUTCOME MEASURES:

1. Primary Outcome: Summary of Adverse Events Reported in Participants That Received a Single Intramuscular Dose of Adacel™
Description: All adverse event reported by vaccinated subjects within 30 days post-vaccination during the 6 year post marketing surveillance period.
Time Frame: 30 days post-vaccination
Population: Safety events were assessed in the Safety Analysis Set.
Measure: Number; unit: Participants
Arm/Group | Study Subjects
Number analyzed (Participants) | 659
Participants
  Adverse events | 168
  Serious adverse events | 1
  Unexpected adverse events | 68

2. Other Pre Specified Outcome: Number of Participants Reporting Unexpected Adverse Events After A Single Intramuscular Dose of Adacel™
Description: Unexpected adverse events reported by vaccinated subjects within 30 days post-vaccination during the 6 year post marketing surveillance period.
Time Frame: 30 days post-vaccination
Population: Safety events were assessed in the Safety Analysis Set.
Measure: Number; unit: Participants
Arm/Group | Study Subjects
Number analyzed (Participants) | 659
Participants
  Myalgia | 26
  Bronchitis | 11
  Rhinitis | 6
  Coughing | 3
  Rhinorrhoea | 3
  Nasopharyngitis | 2
  Pharyngitis | 2
  Throat sore | 2
  Asthma | 1
  Nasal obstruction | 1
  Sputum | 1
  Tonsillitis | 1
  Malaise | 14
  Influenza | 2
  Pain axillary | 1
  Purulent discharge | 1
  Gastritis | 8
  Gastritis acute | 3
  Gastroenteritis | 3
  Enteritis | 2
  Dyspepsia | 1
  Dermatitis atopic | 1
  Furuncle (excluding genital) | 1
  Rash impetiginous | 1
  Sweating increased | 1
  Dizziness | 3
  Allergic conjunctivitis | 1
  Conjunctivitis | 1
  ALT increased | 1
  AST increased | 1
  Hand foot mouth disease | 1

3. Other Pre Specified Outcome: Number of Participants Reporting Adverse Events After A Single Intramuscular Dose of Adacel™
Description: as for outcome 1
Time Frame: 30 days post-vaccination
Population: Safety events were assessed in the Safety Analysis Set.
Measure: Number; unit: Participants
Arm/Group | Study Subjects
Number analyzed (Participants) | 659
Participants
  Injection-site Pain | 108
  Injection-site Erythema | 46
  Injection-site Swelling | 42
  Injection-site Itching | 5
  Injection-site Bruising | 1
  Myalgia | 26
  Arthralgia | 1
  Bronchitis | 11
  Rhinitis | 6
  Coughing | 3
  Rhinorrhoea | 3
  Nasopharyngitis | 2
  Pharyngitis | 2
  Throat sore | 2
  Asthma | 1
  Nasal obstruction | 1
  Sputum | 1
  Tonsillitis | 1
  Malaise | 14
  Fever | 7
  Influenza | 2
  Knee pain | 1
  Pain axillary | 1
  Purulent discharge | 1
  Gastritis | 8
  Gastritis acute | 3
  Gastroenteritis | 3
  Diarrhoea | 2
  Enteritis | 2
  Dyspepsia | 1
  Nausea | 1
  Vomiting | 1
  Headache | 13
  Dizziness | 3
  Dermatitis atopic | 1
  Furuncle (excluding genital) | 1
  Itching | 1
  Rash | 1
  Rash impetiginous | 1
  Sweating increased | 1
  Allergic conjunctivitis | 1
  Conjunctivitis | 1
  ALT increased | 1
  AST increased | 1
  Hand foot and mouth disease | 1

4. Other Pre Specified Outcome: Number of Reported Solicited Injection-Site and Systemic Events Following A Single Intramuscular Dose of Adacel™
Description: Solicited injection-site: Pain, Erythema, and Swelling. Solicited systemic reactions: Fever (Temperature), Headache, Malaise, and Myalgia. Grade 3 Solicited injection-site: Pain, Prevents daily activities; Erythema and Swelling,> 10 cm. Grade 3 Solicited systemic reactions: Fever, ≥39.0°C; Headache, Malaise, and Myalgia, Prevents daily activities.
  All events reported by vaccinated subjects within 7 days post-vaccination during the 6 year post marketing surveillance period.
Time Frame: 7 days post-vaccination
Population: Safety events were assessed in the Safety Analysis Set.
Measure: Number; unit: Number of Events
Arm/Group | Study Subjects
Number analyzed (Participants) | 659
Number of Events
  Any Injection-site Pain | 108
  Grade 3 Injection-site Pain | 0
  Any Injection-site Erythema | 46
  Grade 3 Injection-site Erythema | 0
  Any Injection-site Swelling | 42
  Grade 3 Injection-site Swelling | 1
  Any Fever | 4
  Grade 3 Fever | 1
  Any Headache | 12
  Grade 3 Headache | 0
  Any Malaise | 14
  Grade 3 Malaise | 1
  Any Myalgia | 24
  Grade 3 Myalgia | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected within 30 days of each vaccination during the 6 years post marketing surveillance period.
Arm/Group | Study Subjects
Serious Adverse Events (participants affected / at risk) | 1/659
Other Adverse Events (participants affected / at risk) | 108/659
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Subjects (N=659)
Knee pain (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.00% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Study Subjects (N=659)
Injection-site Pain (General disorders) | 108 (108)
Injection-site Erythema (General disorders) | 46 (46)
Injection-site Swelling (General disorders) | 42 (42)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications